CLINICAL TRIAL: NCT01200160
Title: Post-Marketing Observational Study on the Effectiveness and Safety of Niaspan® in the Treatment of Lipid Abnormalities in Latin America
Brief Title: Study of the Effectiveness and Safety of Niaspan ® in the Treatment of Lipid Abnormalities in Latin America
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: QUASY (Unknown)
Responsible Party: Sponsor
Other Study IDs: P12-055
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-05

CONDITIONS: Cardiovascular Diseases
Keywords: Low-Density Lipoprotein Cholesterol; Hypertriglyceridemia; Latin America; Cardiovascular Diseases; Cholesterol; Sedentary Lifestyle; High-Density Lipoprotein Cholesterol
MeSH Terms: conditions — Cardiovascular Diseases; Hypertriglyceridemia; Sedentary Behavior | interventions — Niacin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Lipid abnormalities: Niacin
  Interventions: Drug: Niacin

INTERVENTIONS:
Drug: Niacin
  Other Names: Niaspan

SUMMARY:
Post-Marketing Observational study of Niaspan® tablet in accordance with each country regulations. This study will be conducted in a prospective, single-arm, multi-center format. As this study is observational in nature, the follow-up of subject's is not prescriptive in nature and is according to the judgment of the physician (investigator in the course of treatment for each patient), within the period of observation of 12 months. This includes an enrollment period of 6 months in which each subject will be observed for approximately 6 months. Examinations, diagnostic measures, findings and observations performed as per usual medical practice during the observation period will be recorded on Case Report Forms (CRFs) by the investigator or site staffs according to the protocol.

DETAILED DESCRIPTION:
This is a Post-Marketing Observational study (PMOS) of Niaspan® tablet in accordance with each country regulations. This study will be conducted in a prospective, single-arm, multi-center format. As this study is observational in nature, the follow-up of subject's is not prescriptive in nature and is according to the judgment of the physician (investigator in the course of treatment for each patient), within the period of 12 months. This includes an enrollment period of 6 months and a treatment duration in which each subject will be observed for approximately 6 months. Examinations, diagnostic measures, findings and observations performed as per usual medical practice during the observation period will be recorded on CRFs by the investigator or site staffs according to the protocol.

Prior to enrollment in the study, each subject will be required to give their written informed consent to participate in the study. Written informed consent will include a statement authorizing the use and/or disclosure of their personal and/or health data. The subject will be assured that patient confidentiality will be maintained at all times according to the local regulations, and that data that might identify the patient will not be collected

For patient's consenting to participate in this PMOS study and meeting all of the inclusion and none of the exclusion criteria, at the initial visit or baseline as well at subsequent visits if appropriate , their demographic, medical history, physical examination, vital sign, flushing/adverse event assessments, concomitant medication information, Niaspan dose change/compliance, and lab testing will be documented as per standard medical practice in each country, although not in a protocolized manner.

If Niaspan® treatment is discontinued, subjects will be followed for another 1 month for any adverse event.

ELIGIBILITY:
Inclusion Criteria

* Male and female subject >18 years-old
* Subjects with primary hyperlipidemia or mixed dyslipidemia with elevated levels of total cholesterol,, LDL-C (low-density lipoprotein-cholesterol), triglycerides and/or decreased levels of HDL-C (high-density lipoprotein-cholesterol) (< 40 mg/dL) and has demonstrated an inadequate response to a lipid-restricted diet and other non-pharmacologic measures alone such as exercise
* Subject has demonstrated persistent dyslipidemic values and/or inadequate response or intolerance to other pharmacologic therapies such as statins, fibrates, resins, etc.
* Female subjects with reproductive potential must use an approved contraceptive method (intrauterine device (IUD), birth control pills or barrier device) during and for 3 months after discontinuation of study treatment.

Exclusion Criteria

* Subject has been treated with any other investigational product in the last 30 days before the day of the screening visit
* Subject exhibits signs of acute illness with clinically relevant findings in the pre-study examination
* Subject has known hypersensitivity to niacin or any component of Niaspan®
* Subject has significant or unexplained hepatic and/or renal dysfunction
* Subject has active peptic ulcer disease
* Subject exhibits active arterial bleeding
* Subject is pregnant or lactating
* The mental condition of the subject renders him/her unable to understand the nature, scope, and possible consequences of the study
* Subject is unlikely to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2010-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique C Morales Villegas, MD, Principal Investigator — Centro de Investigación Cardiometabólica
Locations (22):
- Colombia (2):
  - Site Reference ID/Investigator# 48183, Cali
  - Site Reference ID/Investigator# 48182, Cali
- Mexico (15):
  - Site Reference ID/Investigator# 42108, Aguascalientes
  - Site Reference ID/Investigator# 42110, Aguascalientes
  - Site Reference ID/Investigator# 42103, Guadalajara, Jalisco
  - Site Reference ID/Investigator# 42105, Metepec, Estado de Mexico
  - Site Reference ID/Investigator# 26348, Mexico City
  - Site Reference ID/Investigator# 42102, Mexico City DF
  - Site Reference ID/Investigator# 42107, Mexico City DF
  - Site Reference ID/Investigator# 42109, Mexico City DF
  - Site Reference ID/Investigator# 42106, Mexico City DF
  - Site Reference ID/Investigator# 42104, Tijuana, Baja California Norte
  - Site Reference ID/Investigator# 42112, Tijuana, Baja California Norte
  - Site Reference ID/Investigator# 42111, Tuxtla Gutierrez, Chiapas
  - Site Reference ID/Investigator# 42114, Tuxtla Gutierrez, Chiapas
  - Site Reference ID/Investigator# 42113, Zacatecas City
  - Site Reference ID/Investigator# 42115, Zapopan, Jalisco
- Venezuela (5):
  - Site Reference ID/Investigator# 44202, Bolívar
  - Site Reference ID/Investigator# 26350, Caracas
  - Site Reference ID/Investigator# 44206, Caracas
  - Site Reference ID/Investigator# 44203, Caracas
  - Site Reference ID/Investigator# 44204, Estado Carabobo

RESULTS

PARTICIPANT FLOW:
Groups:
- Lipid Abnormalities: No comparison groups for this observational study. Patients receive only one type of formulation, then drug exposure was the same for all patients.
  This study was conducted in a prospective, single-arm, multi-center format. As this study was observational in nature, the follow-up of subject's was not prescriptive in nature and was according to the judgment of the investigator, within the period of observation set forth in the protocol.
  Typically, Niaspan is titrated in the following manner: After Week 8, titrate to patient response and tolerance. If response to 1000 mg daily is inadequate increase dose to 1500 mg daily; may subsequently increase dose to 2000 mg daily. Ideally, Niaspan should not be increased more than 500 mg in a 4-week period and daily doses above 2000 mg are not recommended. It is expected that women may respond at lower doses than men. However, consult with the approved label for titration recommendation in the particular country.
Period: Overall Study
Arm/Group | Lipid Abnormalities
Started | 128
Completed | 66
Not Completed | 62

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT) population defined as all enrolled subjects who received at least one dose of study medication
Arm/Group | Lipid Abnormalities
Number analyzed (Participants) | 128
Age, Categorical [Number; unit: participants] — There were 128 recruited patients, however for one patient information about birth date is missing, then age is not possible to be calculated. Then descriptive data for "age" is for 127 patients.
  participants
    <=18 years | 0
    Between 18 and 65 years | 96
    >=65 years | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 75
Region of Enrollment [Number; unit: participants]
  Mexico | 53
  Venezuela | 60
  Colombia | 15

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Niaspan
Description: Increasing serum HDL-C (high-density lipoprotein - cholesterol) levels.
  Calculated change in different variables (Difference percent for HDL, LDL, Non-HDL and Triglycerides) was obtained using the expression:
  percent.change=((final.visit.variable-baseline.variable.))/(baseline.variable))*100 Then percent change is calculated at 24 weeks regarding baseline for different variables.
Time Frame: 24 weeks regarding baseline visit (visit1)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HDL-Cholesterol
Number analyzed (Participants) | 53
mg/dL | 41.9755 (7.56248)

2. Secondary Outcome: Evaluate Changes Induced by Niaspan at the Completion of the Study Against Base Line Values
Description: Evaluation of changes in non-HDL-C (non-high-density lipoproteins-cholesterol) lipids, LDL- C (low-density lipoproteins-cholesterol), total cholesterol and triglycerides (including in subjects with high triglycerides ≥ 200 mg/dL), and the impact on the Framingham score
Time Frame: every 4 to 8 weeks for 24 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Frequency of Flushing Events
Description: evaluate occurrence of such events over time
Time Frame: every 4 weeks for 24 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Overall Safety and Tolerability of Niaspan
Description: Evaluate overall safety of Niaspan through evaluation of adverse events
Time Frame: every 4 weeks for 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 weeks
Groups:
- Lipid Abnormalities: Those with the condition and exposed to the study drug
Arm/Group | Lipid Abnormalities
Serious Adverse Events (participants affected / at risk) | 0/128
Other Adverse Events (participants affected / at risk) | 31/128
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lipid Abnormalities (N=128)
Flushing (Skin and subcutaneous tissue disorders) | 31 (35)

LIMITATIONS AND CAVEATS:
Expected sample size was not achieved due to supply issues with the new formulation in Mexico and the local decision in Colombia to cancel marketing the product in the country.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An agreement is in place that includes a clause of keeping Abbott´s information confidential and that any publication would be performed under agreement with Abbott.